CLINICAL TRIAL: NCT01454674
Title: The Vegetable Dose Response Study: Effects of Consumption on Inflammation and Oxidative Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Julie West, Study coordinator, University of Arizona
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 07-0820-02
Record Dates: First submitted 2011-08-11; First posted 2011-10-19 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: 2, 5 & 10 Vegetable doses — 2,5 & 10 serving dose/day combination of fresh lettuce mix, baby carrots, red bell peppers & tomatoes consumed for 3 week intervals

SUMMARY:
The investigators have designed a three dose level, cross-over vegetable feeding study using expertise from nutritional sciences and plant sciences to:

1. Implement a randomized vegetable feeding trial among overweight post- menopausal women
2. Produce, in a controlled environmental setting, vegetable crops which provide a selected variety and quantity of carotenoid and nutrient exposure
3. Assess changes and hopefully demonstrate a significant reduction in oxidant stress and inflammation in this population at risk for developing chronic disease

DETAILED DESCRIPTION:
Women were randomly assigned a vegetable feeding dose order of consuming 2,5 & 10 servings/day of vegetables for 3 week periods, with feeding periods separated by 4 week washout periods, during which time a limited number of low biological value fruits and vegetables were eaten.

This research will provide important and relevant information to fill several gaps in our current knowledge including a more thorough description of the oxidant stress and inflammatory status of overweight, postmenopausal women, assessment of the relevant daily "dose" of vegetables necessary to modulate biomarkers of oxidant stress and inflammation in overweight postmenopausal women and evaluation of the association between plasma nutrient and carotenoid levels in relation to changes in oxidant stress and inflammation in this population. Our long-term goal is to reduce chronic disease risk among "at-risk" post-menopausal females.

ELIGIBILITY:
Inclusion Criteria:

1. Female;
2. Age 50 to 75 years of age;
3. Target to include 20% minority subjects.
4. Post-menopausal - defined as greater than 12 months without menses; or lab values indicative of post-menopausal status;
5. Waist to hip ratio of > 0.85;
6. Body mass index (BMI) between 25.0 and 45 kg/m2 ;
7. Non-smoker;
8. Reported alcohol intake of < 2 servings daily;
9. Reported stable body weight for previous 6 months;
10. In general good health with no history of cancer (other than non- melanoma skin cancer), diabetes, liver or renal disease;
11. No known allergies to or intolerances of leaf lettuce, tomato, carrots or peppers;
12. Willing and able to successfully complete run-in activities -

Exclusion Criteria:

1. Morbid obesity (BMI > 45 kg/m2);
2. Medical diagnosis requiring a therapeutic diet (i.e, diabetes, hepatic disease, etc);
3. Smoking history within previous 6 months;
4. Consuming > 5 servings of fruits/vegetables daily prior to study enrollment;
5. Regular use of anti-inflammatory medications;
6. Unwilling to discontinue dietary supplements with the exception of study provided multivitamin and/or calcium supplement;
7. Unwilling to adhere to study protocol including limiting fruit intake to 1 serving per day and excluding vegetable intake other than study provided and allowed vegetables.
8. Participating in greater than 10 hours of regularly scheduled physical activity weekly or participating in vigorous physical activity on a regular basis (i.e. daily running, contact sports, etc) as assessed using a validated physical activity assessment questionnaire.

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-10; Primary Completion 2010-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Serum high sensitivity c-reactive protein | Change between baseline and 3 weeks
  Change in serum high sensitivity c-reactive protein
Urine Isoprostanes 8-epi-PGF2alpha | Change between baseline and 3 weeks
  Change in Urine Isoprostanes 8-epi-PGF2alpha

SECONDARY OUTCOMES:
Plasma carotenoids | Change between baseline and 3 weeks
  Change in plasma carotenoids.
Physical activity - Arizona Activity Frequency Questionnaire | Change between baseline and 21 weeks
  Change in physical activity.
Body weight | Change between baseline and 3 weeks
  Change in body weight
Waist/hip circumference | Change between baseline and 3 weeks
  Change in waist/hip circumference
Percent body fat | Change between baseline and 3 weeks
  Change in % body fat
Blood pressure | Change between baseline and 21 weeks
  Change in blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Thomson, PhD, RD, Principal Investigator — U of AZ Nutritional Sciences Department
Locations (1):
- U of AZ Nutritional Sciences Department, Tucson, Arizona, United States